CLINICAL TRIAL: NCT04309058
Title: Observation of the Effect of Vitamin D Supplementation on Chronic Course of Patients With Ulcerative Colitis Based on Vitamin D Receptor Fok I Gene Polymorphism,a Prospective Cohort Study
Brief Title: Observation of the Effect of Vitamin D Supplementation on Chronic Course of Patients With Ulcerative Colitis Based on Vitamin D Receptor Fok I Gene Polymorphism
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2017-01-121
Record Dates: First submitted 2020-02-24; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Ulcerative Colitis; Vitamin D Deficiency; Vitamin D Supplement
MeSH Terms: conditions — Colitis, Ulcerative; Vitamin D Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D drops (Experimental): This group of patients are going to supplemented with Vitamin D drops 400IU / d orally.
  Interventions: Drug: Vitamin D drops
- Control (No Intervention): The other group do not interfere.

INTERVENTIONS:
Drug: Vitamin D drops — Vitamin D-deficient UC patients are divided into two groups, one group is given orally with Vitamin D drops 400IU / d, while the other group do not interfere.
  Arms: Vitamin D drops

SUMMARY:
Aims:Prospectively observe the effects of Vitamin D drops supplementation on the chronic course of ulcerative colitis patients, analyze whether the effect of Vitamin D drops on UC patients is affected by factors such as disease site, disease activity, treatment, etc.Exploring the relationship between Fok I gene polymorphism and the efficacy of vitamin D supplementation. Provide a certain theoretical basis for "precision treatment" for UC patients in the future.

Design：It is a prospective cohort study. Investigators include a total of 100 participants with UC according to the inclusion and exclusion criteria, and divide them into two groups to assess their initial disease activity and detect related indicators. At the same time，investigators detect the Fok I gene polymorphism in all participants.One group is given Vitamin D drops 400IU per day orally, and the control group do not intervene. Participants' disease activity is assessed at baseline and related indicators are determined. The disease activity is re-evaluated in the 3rd, 6th, 9th, and 12th months, and the serum indexes are re-evaluated.Investigators use statistical methods to analyze whether Vitamin D drops supplementation treatment can increase the serum 25 (OH) D level of UC participants, improve the condition of UC participants,relationship with Fok I gene polymorphism，and analyze the effects of Vitamin D drops on participants with UC is affected by factors such as disease site, disease activity, and treatment.

DETAILED DESCRIPTION:
1. The research can be started only after approval by the Medical Ethics Committee of the Second Affiliated Hospital of Wenzhou Medical University.
2. According to the "Consensus on Diagnosis and Treatment of Inflammatory Bowel Disease" formulated by the Beijing Conference in 2018 as a standard, patients with clear diagnosis of UC are collected.Other diagnostic criteria include Vitamin D deficiency (<= 20ng / ml). Exclusion criteria included pregnancy, breastfeeding, liver and kidney dysfunction, concurrent autoimmune diseases, and use of antiepileptic drugs or drugs metabolized by liver cytochrome P450 enzymes.
3. Assess disease activity of UC participants based on the "Moya score".
4. General information about participants with UC is collected.
5. Detection of Fok I gene polymorphism using Snapshot technology.
6. The level of serum 25 (OH) D of participants is detected.
7. Serum C-reactive protein, erythrocyte sedimentation rate, albumin, calcium and phosphorus levels are measured.
8. Develop a treatment plan for all participants.
9. Participants are divided into two groups, one group is given oral Vitamin D drops 400IU/ d, and the other group do not intervene.
10. The disease activity is re-evaluated in the 3rd, 6th, 9th, and 12th months, and the above serum indexes are re-evaluated.
11. Follow-up for 12 months. By comparing the above indicators, observe that in the Han population:

    1. Can Vitamin D drops supplementation increase serum 25 (OH) D levels in patients with UC?
    2. Can Vitamin D drops supplementation improve the condition of patients with UC?
    3. Whether Fok I gene polymorphism affect the efficacy of Vitamin D drops supplementation therapy?
    4. Whether the effects of Vitamin D drops on UC patients is affected by factors such as disease site, disease activity, treatment, etc ..
12. Through statistical analysis, comprehensive analysis of the effectiveness and safety of Vitamin D drops supplementation in Han patients with UC, and its relationship with Fok I gene polymorphism, providing a theoretical basis for further "precise treatment" intervention in inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Clearly diagnosed patients with UC
* Vitamin D deficiency (<= 20ng / ml)

Exclusion Criteria:

* Pregnancy, lactation
* Liver and kidney insufficiency
* Co-morbid with other autoimmune diseases
* Use antiepileptic drugs or drugs metabolized by liver cytochrome P450 enzymes
* Vitamin D level is normal or high

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Genotype frequency of vitamin D receptor single nucleotide polymorphisms in participants | 1 year
  Genotype frequency of vitamin D receptor single nucleotide polymorphisms in participants can reflect whether it is related to the severity of the disease and how much relevance.
Serum 25 (OH) D level | 1year
  Because serum 25 (OH) D levels are relatively stable, they are considered the most reliable indicator of vitamin D status

SECONDARY OUTCOMES:
Blood calcium and phosphorus | 1year
  Monitoring serum calcium and phosphorus levels to prevent toxic side effects.
erythrocyte sedimentation rate | 1year
  ESR can be used to reflect the degree of inflammation in the body.
Concentration of C-reactive protein in participants | 1year
  Concentration of C-reactive protein can be used to reflect the degree of inflammation in the human body.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang yi, PhD, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- SAHWenzhouMU, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Data sets will be made available on relevant requests and in accordance with journal guidelines when publishing results from this study.